CLINICAL TRIAL: NCT06037018
Title: A Phase 1 Study to Evaluate the Safety, Pharmacokinetics, Pharmacodynamics, and Preliminary Anti-tumor Efficacy of CC312 in Adult Patients With Relapsed/Refractory CD19 Positive B-cell Hematologic Malignancies
Brief Title: Safety Study of CC312 in Adult Patients With Relapsed/Refractory CD19 Positive B-cell Hematologic Malignancies
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: CytoCares Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CC312-001(C)
Record Dates: First submitted 2023-08-28; First posted 2023-09-14 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Non-hodgkin Lymphoma; Acute Lymphoblastic Leukaemia; Chronic Lymphocytic Leukemia
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Lymphocytic, Chronic, B-Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CC312 (Experimental)
  Interventions: Biological: CC312

INTERVENTIONS:
Biological: CC312 — Doses from 0.3 to 45 µg/dose by intravenous infusion

SUMMARY:
This is a Phase 1, open-label, dose-escalation study to evaluate the safety, PK, PD and immunogenicity of CC312 following intravenous doses of CC312 in patients with relapsed and refractory (r/r) CD19 expressing B-cell non-Hodgkin lymphoma and B-cell lymphocytic leukemia.

DETAILED DESCRIPTION:
This study is an accelerated dose titration design divided into 2 parts.

Part 1 of the study is an accelerated dose-escalation design involving 5 dose levels: 0.3, 0.6, 1.2, 2.4 and 4.8 mcg given intravenously (IV) with cohorts of one patient per dose level. Patients in this part will receive 1 priming dose (D-7) and 1 intermediate dose of CC312 (D-3) on the first week, followed by twice weekly dosing of escalated dose for three weeks beginning on the second week. The dose limiting toxicity (DLT) observation period will be 28 days. The optimal priming dose and intermediate dose level will be determined in this part.

Part 2-A will follow a standard 3 + 3 dose escalation design using five dose levels: 9.6, 16, 24, 34 and 45 μg to obtain data on the safety and tolerability of CC312. Patients in this part will receive priming dose and intermediate dose of CC312 established in Part 1 before given the treatment dose. MTD or RP2D will be determined in Part 2-A and tested in expanded population(Part 2-B).

Part 2-B is planned for cohorts of 6-10 patients with B-cell non-Hodgkin lymphoma or B-cell lymphocytic leukemia receiving priming/ treatment dose levels as defined in the Part 1 and Part 2-A study.

ELIGIBILITY:
Inclusion Criteria:

1. CD19 positive B-cell malignancies confirmed as one of the following: aggressive or indolent B-cell NHL, philadelphia chromosome-positive or -negative B-cell ALL, or B-cell CLL; patient must meet the definition of relapse/refractory before enrollment.
2. ECOG (Eastern Cooperative Oncology Group) performance status 0-2, life expectancy >3 months；
3. Clinical laboratory values as specified below during the Screening period.

   * Total bilirubin <1.5 ULN, may be elevated up to 3 x ULN if the elevation can be reasonably ascribed to the presence of metastatic disease in the liver or in patients with documented Gilbert's Syndrome;
   * ALT or AST <3ULN, may be elevated up to 5 x ULN if the elevation can be reasonably ascribed to the presence of metastatic disease in liver;
   * Calculated creatinine clearance > 50 mL/min (The Cockcroft-Gault formula);
   * Hemoglobin ≥ 7 g/dL;
   * Neutrophil count > 1,000/mm3 for B-cell NHL patient;
   * Platelet count > 75,000/mm3 for B-cell NHL patient;
   * B-ALL patients must have peripheral blast count ≤ 30,000/ mm3 prior to first dose of CC312.
   * Prothrombin time-international normalized ratio (PT-INR) ≤ 1.5ULN.
4. Female patients of childbearing potential or male patients with a partner of childbearing potential must use one or more contraception methods from screening and continued during study treatment until 3 months after the last dose;
5. Ability to understand and willingness to provide written informed consent and to comply with scheduled visits and study procedures.

Exclusion Criteria:

1. Systemic anticancer therapy within 5 half-lives of the agent or attending clinical trials 4 weeks prior to beginning CC312;
2. Treatment with radiotherapy within 2 weeks before the study entry;
3. Treatment with CAR-T within 3 months before the study entry;
4. Active serious infection requiring antibiotics within 14 days before study entry;
5. Patients with prior treatment with anti-CD19 directed therapies are eligible only if their tumor cells have been shown to express CD19 after completing the CD19-directed therapy;
6. Patients with brain metastases or other significant neurological conditions, except for brain metastases which are asymptomatic and radiologically stable without need for steroids for 2 weeks before the first dose of CC312;
7. Treatment with corticosteroids (>10mg daily prednisone or equivalent) or immunosuppressive medication ≤ 7 days before the first dose of CC312, with the following exceptions:

   * Topical, ocular, intra-articular, intranasal, or inhalational corticosteroids;
   * Use of dexamethasone to reduce peripheral blast counts in ALL;
8. Vaccination with a live virus vaccine within 4 weeks prior to the study enrollment;
9. Current autoimmune disease or history of autoimmune disease with potential CNS involvement;
10. Known to be allergic to protein drugs or recombinant proteins or excipients in the CC312 drug formulation. Patients who experienced Grade 3 reactions that lasted < 24h may be eligible after discussion with investigator；
11. Except for the tolerable events determined by the investigator, any toxic effects of the prior therapy which have not resolved to Grade 1 (CTCAE v5.0);
12. Admission or evidence of illicit drug use, drug abuse, or alcohol abuse;
13. Cerebrovascular accident (CVA), Transient ischemic attack (TIA), myocardial infarction (MI), unstable angina, or New York Heart Association (NYHA) class III or IV heart failure occurring within <6 months of study entry; uncontrolled arrhythmia within < 3 months of study entry. Patients with rate-controlled arrhythmias may be eligible for study entry at discretion of the Investigator.;
14. Major surgery < 4 weeks or minor surgery < 2 weeks prior to screening; wound must be fully healed (minor surgical procedures such as catheter placement are not exclusionary criteria);
15. Existence of congenital long QT syndrome, QTcF > 450 msec (for male) or 470 msec (for female), use of cardiac pacemaker, left ventricular ejection fraction (LVEF) <50%, clinically significant arrhythmia that requires intervention, cardiac troponin I or T > 2.0 ULN, poorly controlled diabetes (HbA1c > 9%), hypertension (systolic pressure > 160 mmHg or diastolic pressure > 100mmHg), or other medical conditions as determined by the Investigator. Patients with stable atrial fibrillation or flutter are eligible for study entry at the discretion of the Investigator;
16. Any other serious underlying medical (e.g. active gastric ulcer, uncontrolled seizures, cerebrovascular incidents, gastrointestinal bleeding, severe signs and symptoms of coagulation and clotting disorders, cardiac conditions), psychiatric, psychological, familial or geographical condition that, in the judgment of the Investigator, may interfere with the planned staging, treatment and follow-up, affect patient compliance or place the patient at high risk for treatmentrelated complications;
17. Concurrent malignancy < 5 years prior to entry other than adequately treated cervical carcinoma-in-situ, localized squamous cell cancer of the skin, basal cell carcinoma, localized prostate cancer, ductal carcinoma in situ of the breast, or < T1 urothelial carcinoma. Patients with prostate cancer that is under active surveillance are eligible.;
18. Pregnant or nursing women.;
19. Active hepatitis B：HBsAg positive and HBV-DNA>ULN; Active hepatitis C：HCV-Ab positive and HCV-RNA>ULN；
20. Known HIV infection；
21. B-NHL patient that received autologous stem cell transplant 6 months prior to study screening, or historically received organ or allogeneic stem cell/bone marrow transplant;
22. B-ALL patients that received transplantation treatment within 3 months prior to enrollment in the study.;
23. Subjects who in the judgement of the Investigator are not suited to participate in this trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2023-08-07 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Dose limiting toxicities (DLTs) | From the first infusion of CC312 till the end of the 28 days DLT（Dose Limiting Toxicity）observation period.
  Toxicity will be evaluated according to the NCI CTCAE, Version 5.0, except CRS which will be graded according to ASTCT Consensus Grading for CRS.
Incidence and severity of adverse event (AE) | From the first infusion of CC312 until 28 days following the end of treatment.
  Overall numbers of participants with any AE, including any laboratory abnormality, treatment-emergent adverse event (TEAE), and serious adverse events (SAE). Severity (toxicity grade) for each AE will be determined using the NCI CTCAE, version 5.0; except cytokine release syndrom (CRS) and immune effector cell-associated neurotoxicity syndrome (ICANS) which will be graded according to ASTCT Consensus Grading.

SECONDARY OUTCOMES:
Pharmacokinetics (PK): serum concentration | Cycle 1: baseline (Day -10~Day -8); 1 hour-pre-dose and multiple-timepoints-post-dose; Cycle 2 and subsequent cycle: 1 hour-pre-dose; after the end of treatment (EOT)/withdraw/at the end of study (EOS). Length of each cycle: 28 days.
  Blood samples will be collected to analysis serum concentration of CC312. Derived PK parameters will be calculated using the non-compartmental model.
Pharmacodynamics (PD): cytokine analysis | Cycle 1: baseline (Day -10~Day -8); 1 hour-pre-dose and multiple-timepoints-post-dose; Cycle 2 and subsequent cycle: 1 hour-pre-dose; after the end of treatment (EOT)/withdraw/at the end of study (EOS). Length of each cycle: 28 days.
  Peripheral blood will be collected for CRS-related cytokine analysis in all dose escalation cohorts.
Pharmacodynamics (PD): immunophenotyping | Cycle 1: baseline (Day -10~Day -8); 1 hour-pre-dose and multiple-timepoints-post-dose; Cycle 2 and subsequent cycle: 1 hour-pre-dose; after the end of treatment (EOT)/withdraw/at the end of study (EOS). Length of each cycle: 28 days.
  Peripheral blood will be collected for immunophenotyping (including the activation of CD4+ and CD8+ T cells, and depletion of B cells) in all dose escalation cohorts.
Immunogenicity: anti-CC312 antibody | Cycle 1: baseline (Day -10~Day -8); 1 hour-pre-dose on Day-7/Day 8. Cycle 2 and subsequent cycle: within 1 hour before infusion on Day 1/Day 15; after the end of treatment (EOT)/withdraw/at the end of study (EOS). Length of each cycle: 28 days.
  The proportions of participants with positive anti-drug antibody (ADA) status and those with positive neutralizing anti-drug antibody (NAb) status will be presented by descriptive statistics.

OTHER OUTCOMES:
Tumor response to CC312 | From the first infusion of CC312 until 28 days following the end of treatment.
  B-NHL, B-ALL and CLL will be evaluated by Lugano criteria, NCCN Guidelines 2021, and iwCLL guidelines 2008, respectively. Therapeutic endpoints includes: overall response rate [ORR] (including complete remission [CR] and partial remission [PR]), duration of overall response [DOR], disease control rate [DCR], and relapse-free survival [RFS] in participants.

CONTACTS AND LOCATIONS:
Overall Officials: JUNYUAN QI, MD, Principal Investigator — Institute of Hematology & Blood Diseases Hospital, China
Locations (1):
- InstituteHBDH, Tianjin, Tianjin Municipality, China